CLINICAL TRIAL: NCT01923493
Title: Chronic Neck Pain: a Randomized Controlled Trial in Patients With Chronic Neck Pain Comparing Tuina vs. no Intervention Waiting List
Brief Title: Tuina for Patients With Chronic Neck Pain
Acronym: tuina
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Claudia M. Witt, Prof. Dr. med., Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Tuina-13
Record Dates: First submitted 2013-08-13; First posted 2013-08-15 (Estimated); Last update posted 2015-02-09 (Estimated); Status verified 2015-02

CONDITIONS: Chronic Neck Pain
Keywords: neck pain; tuina
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- no intervention waiting list (Active Comparator): Patients in the no intervention waiting list group will not receive a study intervention.
  Interventions: Other: no intervention
- tuina (Experimental): tuina treatment
  Interventions: Other: tuina

INTERVENTIONS:
Other: tuina — Patients in the tuina group will receive a tuina therapy (also known as Chinese massage). A Chinese massage lasts about 20 to 30 minutes. A series of 6 sessions with 2 treatments per week is applied.
  Other Names: chinese massage
  Arms: tuina
Other: no intervention — Patients in the no intervention waiting list group will not receive a study intervention. They will continue their respective pre-study therapy during the study period.
  Arms: no intervention waiting list

SUMMARY:
The aim is to evaluate whether tuina is more effective and cost-effective than no intervention waiting list to reduce neck pain measured on a visual analogue scale in patients suffering from chronic neck pain.

DETAILED DESCRIPTION:
Objective: To evaluate whether tuina is more effective and cost-effective than no intervention waiting list to reduce neck pain measured on a visual analogue scale in patients suffering from chronic neck pain.

Study Design: Open single-centre randomized two-armed controlled trial. Setting: The study will be performed at a University out-patient clinic specialized in Integrative Medicine, with experience in the treatment of chronic pain.

Participants: 88 outpatients with chronic neck pain, who will be randomly allocated to two groups (tuina, or no intervention (control)).

Intervention: Patients receive either six tuina treatments within 3 weeks or no additional intervention.

Main outcome measure: The primary outcome is the mean neck pain intensity over the last seven days on a visual analogue scale (Huskisson, 1974) (VAS, 0-100 mm, 0 = no pain, 100= worst imaginable pain) after four weeks.

ELIGIBILITY:
Inclusion Criteria:

* female or male
* 18 to 60 years of age
* clinical diagnosis "chronic neck pain", i.e. neck pain for at least 12 weeks
* if additional back pain is reported, neck pain has to be predominant
* intensity of the average neck pain over the last 7 days had to be more than 40 mm on a 100-mm visual analogue scale (VAS)
* ability to give oral and signed written informed consent
* patient's mental and physical ability to participate in the trial
* willingness to be randomized, to attend visits, to complete questionnaires
* written and oral informed consent

Exclusion Criteria:

* neck pain caused by a malignant disease
* neck pain caused by trauma
* rheumatic disorder
* prior spinal column surgery
* neurological symptoms, e.g. radicular symptoms because of a prolapsed vertebral disc
* suspected osteoporosis
* obesity with BMI ≥30 Kg/m2
* known vascular anomaly such as aneurysm
* regular intake of analgesics (>1x per week) because of a additional diseases
* intake of centrally acting analgesics
* current application for a benefit
* pregnancy
* severe acute and or chronic disease which does not allow participation in the therapy
* other limitations which do not allow participation in the therapy
* alcohol or substance abuse
* tuina treatment during the six months before study entry
* participation in another clinical trial during six months before the study and parallel to the study
* anticipated new treatments which have a positive influence on the neck pain such as physiotherapy against neck pain, acupuncture, massage during the study
* no sufficient German language skills

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 92 (Actual)
Dates: Start 2013-08; Primary Completion 2014-04 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
mean neck pain intensity of the last seven days | 4 weeks

SECONDARY OUTCOMES:
mean neck pain intensity of the last seven days | 12 weeks
Neck Pain and Disability Scale (NPDS) | 4 weeks, 12 weeks
Neck Disability Index (NDI) | 4 weeks, 12 weeks
SF-12 health related quality of life | 4 weeks, 12 weeks
Costs | 4 weeks, 12 weeks
  Data on Resource-consumption and associated costs are planned to be derived as patient-reported information using the patient questionnaires.
Body efficacy expectation | 4 weeks, 12 weeks
  Body-Efficacy Expectation (BEE) is a scale to measure the conviction that one's body is able to deal with health-threatening factors by itself. It is a six items' scale developed in the Institute of Social Medicine, Epidemiology and Health Economics
medication intake | 4 weeks, 12 weeks
  number and type of medication used
number of serious adverse events | 4 weeks, 12 weeks
adverse reactions | 4 weeks, 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Claudia M Witt, MD, Principal Investigator — Institute for Social Medicine, Epidemiology and Health Economics, Charité - Universitätsmedizin Berlin
Locations (1):
- Institute for Social Medicine, Epidemiology and Health Economics Charité Universitätsmedizin Berlin, Berlin, State of Berlin, Germany